CLINICAL TRIAL: NCT03334084
Title: A Randomized, Open-label, Parallel Group Study to Compare the Pharmacokinetics, Pharmacodynamics and Safety and Tolerability of a Subcutaneous Formulation With an Intravenous Formulation of ARGX-113 in Healthy Male Subjects
Brief Title: A Study to Compare the PK, PD and Safety and Tolerability of a SC With an IV Formulation of ARGX-113 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: ARGX-113-1702
Record Dates: First submitted 2017-10-23; First posted 2017-11-07 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Bioavailability Study
MeSH Terms: interventions — efgartigimod alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Experimental): Scheme 1
  Interventions: Drug: ARGX-113
- 2 (Experimental): Scheme 2
  Interventions: Drug: ARGX-113
- 3 (Experimental): Scheme 3
  Interventions: Drug: ARGX-113

INTERVENTIONS:
Drug: ARGX-113 — intravenous or subcutaneous administration

SUMMARY:
The study is a Randomized, Open-label, Parallel Group Study to Compare the Pharmacokinetics, Pharmacodynamics and Safety and Tolerability of a Subcutaneous Formulation With an Intravenous Formulation of ARGX-113 in Healthy Male Subjects

ELIGIBILITY:
Inclusion Criteria:

1. Male, between 18-55 years of age.
2. Body mass index (BMI) between 18-30 kg/m2.
3. Willingness and ability to understand the purpose and risks of the study and provide signed and dated informed consent.
4. Non-vasectomized male subjects having a female partner of childbearing potential must agree to the use of an effective method of contraception until 90 days after the last administration of study drug.
5. Subjects have to agree not to donate sperm until 90 days after the last administration of study drug.
6. Judged by the investigator to be in good health based upon the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and laboratory findings.
7. Agree to discontinue and refrain from intake of all medications, except occasional paracetamol use (maximum dose of 2 g/day and maximum of 10 g/2 weeks), at least 2 weeks prior to the first study drug administration. In addition, subjects must agree to the prohibitions and restrictions for this study.
8. Subject is a non-smoker, and not using any nicotine containing products. A non-smoker is defined as an individual who has abstained from smoking for at least 1 year prior to Screening.

Exclusion Criteria:

1. Known hypersensitivity to study drug ingredients or a significant allergic reaction to any drug as determined by the investigator, such as anaphylaxis requiring hospitalization.
2. Active infection; a recent serious infection (i.e., requiring injectable antimicrobial therapy or hospitalization) within the 8 weeks prior to screening.
3. Subjects with known clinically relevant immunological disorders.
4. History of severe allergic or anaphylactic reactions.
5. Known history or any symptom of clinically significant illness in the 6 months before the first study drug administration.
6. Presence or having sequelae of gastrointestinal, liver, kidney or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
7. History of malignancy within the past 5 years (except for basal cell carcinoma of the skin that has been treated with no evidence of recurrence).
8. Clinically relevant abnormalities detected on ECG regarding either rhythm or conduction (e.g., QTcF > 450 ms [millisecond], or a known long QT syndrome). A first degree heart block or sinus arrhythmia will not be considered as a significant abnormality.
9. Clinically relevant abnormalities detected on vital signs prior to first dosing.
10. Significant blood loss (including blood donation [> 500 mL]), or had a transfusion of any blood product within 12 weeks prior to the initial study drug administration or plan one within 4 weeks after the end of the study.
11. Treatment with any drug known to have a well-defined potential for toxicity to a major organ in the last 3 months preceding the initial study drug administration.
12. The subject has a history of consuming more than 21 units of alcoholic beverages per week or has a history of alcoholism or drug/chemical/substance abuse within past 2 years prior to screening (Note: one unit = 330 mL of beer, 110 mL of wine or 28 mL of spirits).
13. Consumption of a large quantity of coffee, tea (> 6 cups per day) or equivalent.
14. Concurrent participation or participation within 90 days prior to the initial study drug administration in a drug/device or biologic investigational research study.
15. Administration of a vaccine within 60 days prior to initial study drug administration.
16. Administration of any systemic immunosuppressant agent within 6 months prior to initial study drug administration.
17. Administration of any systemic steroid within 2 months prior to initial study drug administration.
18. Administration of an injectable drug within 30 days prior to the initial study drug administration.
19. Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, or other staff or relative thereof who is directly involved in the conduct of the study.
20. Any condition or circumstances that in the opinion of the investigator may make a subject unlikely or unable to complete the study or comply with study procedures and requirements.
21. Unsuitable vein for infusion and/or blood sampling.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2017-10-11 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

PRIMARY OUTCOMES:
bioavailability of a s.c. ARGX-113 formulation | 1.5 months
  AUC0-inf

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Cousin, MD, Study Director — argenx
Locations (1):
- QPS Netherlands B.V., Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No